CLINICAL TRIAL: NCT03341169
Title: Impact of Perioperative Treatment With Intravenous Glutamine on Myocardial Protection in Cardiac Surgery Patients With Aortic Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2017-0774
Record Dates: First submitted 2017-10-23; First posted 2017-11-14 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Aortic Valve Stenois
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-Blinded, Placebo-Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glutamine (Experimental): Intravenous glutamine infusion perioperatively for 18 hours (8 hours before surgery and 10 hours after induction of anesthesia)
  Interventions: Drug: N(2)-L-Alanine L-Glutamine dipeptide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo (0.9% NaCl (normal saline))

INTERVENTIONS:
Drug: N(2)-L-Alanine L-Glutamine dipeptide — :Intravenous infusion of N (2) -L-alanyl-L-glutamine(mixed with normal saline, ratio 1:1) at the dose of 0.25g/kg(body weight) for 8 hours before induction of anesthesia(rate=2.5*weight/8 ml/h) and administration another 0.25g/kg(body weight) of N (2) -L-alanyl-L-glutamine(mixed with 8.5% amino acid solution, ratio 1:5) into the central vein for 10 hours after induction of anesthesia(rate=0.75*weight ml/h)
  Arms: Glutamine
Drug: placebo (0.9% NaCl (normal saline)) — Intravenous infusion of 0.9% NaCl for 8 hours before induction of anesthesia(rate=2.5*weight/8 ml/h) and administration 0.9% NaCl into the central vein for 10 hours after induction of anesthesia(rate=0.75*weight ml/h)
  Arms: Placebo

SUMMARY:
The purpose of this study is to confirm if myocardial protection effect can be obtained by intravenous administration of glutamine in patients undergoing aortic valve replacement with severe aortic stenosis (who are at high risk for ischemia-reperfusion injury). As a prospective double blinded randomized placebo-controlled trial, the investigators detect and compare the degree of myocardial damage(with CK-MB and Troponin T) and myocardial protection (through hsp 70 expression in atrial tissue), cardiovascular index, inflammatory reaction, and clinical manifestation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with between 20 and 80 years scheduled for aortic valve replacement alone or combined surgery including aortic valve replacement due to severe aortic valve stenosis

Exclusion Criteria:

* Patients with renal insufficiency (eGFR 60 ml / min / 1.73 m 2 or less)
* patients who are considering surgery for coronary artery disease or who have a stenosis> 70%
* hemodynamically unstable patients undergoing emergency surgery or patients with intra-aortic balloon pump insertion
* patients unable to make their own decisions, illiterate, foreigners
* epilepsy
* severe metabolic acidosis
* pulmonary edema
* history of myocardial infarction
* elevation of total bilirubin or AST / ALT
* Patients higher than normal, weighing more than 80 kg
* with evidence of infection
* pregnant and lactating women

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-09-28 (Estimated); Study Completion 2019-09-28 (Estimated)

PRIMARY OUTCOMES:
degree of myocardial damage with CK-MB (Creatine Kinase MB lsoenzyme) | 1 day before the operation
degree of myocardial damage with CK-MB (Creatine Kinase MB lsoenzyme) | 10 minutes after ICU(intensive care unit) entrance,
degree of myocardial damage with CK-MB (Creatine Kinase MB lsoenzyme) | 24 hours after surgery
degree of myocardial damage with CK-MB (Creatine Kinase MB lsoenzyme) | 48 hours after surgery
Troponin-T(Tn-T) level | 1 day before the operation
Troponin-T(Tn-T) level | 24 hours after surgery

SECONDARY OUTCOMES:
IL-6 | a day before surgery
IL-6 | 10 minutes after ICU(intensive care unit) entrance
Free fatty acid | a day before surgery
Free fatty acid | 10 minutes after ICU(intensive care unit) entrance
CRP | a day before surgery
CRP | 24 hours after surgery
cardiovascular index | 10 minutes after ICU(intensive care unit) entrance
cardiovascular index | 12 hours after surgery
cardiovascular index | 24 hours after surgery
occurrence of sternal infections | Within 30 days postoperatively
mortality | During hospitalization regardless of length of stay or within 30 days of surgery if discharged
occurrence of cardiovascular complications | up to 1 year
  *cardiovascular (myocardial infarction, heart failure, arrhythmia), cerebral infarction, renal failure: During the hospitalization for surgery, which includes the entire postoperative period up to discharge, even if over 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No